CLINICAL TRIAL: NCT04536662
Title: Comparisons of Different Forms of Glucocorticoid on the Recovery of Reproductive Function in Patients With 21α-hydroxylase Deficiency
Acronym: CGP21
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD-20200819
Record Dates: First submitted 2020-08-23; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone; Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group hydrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone
- Group Prednisone (Experimental)
  Interventions: Drug: Prednisone
- Group Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Hydrocortisone — The initial dose of hydrocortisone (20mg/tablet) was 15mg/m2/day to the maximum dose of 60mg, which was orally administered in three times, with the dose ratio of 2:1:3, and the administration time was 8:00-15:00-21:00.
  Arms: Group hydrocortisone
Drug: Prednisone — The initial dose of prednisone (5mg/tablet) was 3mg/m2/day to the maximum dose of 15mg. The dosage ratio was 1:2 and the administration time was 8:00 and 21:00.
  Arms: Group Prednisone
Drug: Dexamethasone — The initial dose of dexamethasone (0.75mg/tablet) was 0.3mg/m2/day to the maximum dose of 0.75mg and the administration time was 21:00.
  Arms: Group Dexamethasone

SUMMARY:
The purpose of this study is to conduct an open, randomized controlled clinical trial, evaluating the effects of different dosage forms of glucocorticoid on the Recovery of Reproductive Function in Patients With 21α-hydroxylase Deficiency.

DETAILED DESCRIPTION:
In the present study, about 120 patients who are more than 14 years old and diagnosed with 21-hydroxylase deficiency will be enrolled from Ruijin Hospital, Shanghai Jiao Tong University School of Medicine in China. Randomisation was computer generated and stratified by subtype and gender. After screening, eligible subjects will be randomly treated with equivalent dose of hydrocortisone, prednisone or dexamethasone for one year.

The treatment regimen was as follows. Firstly, at least one month washout period (withdrawal) was performed before treatment. The initial dose of hydrocortisone (20mg/tablet) was 15mg/m2/day to the maximum dose of 60mg, which was orally administered in three times, with the dose ratio of 2:1:3, and the administration time was 8:00-15:00-21:00. The initial dose of prednisone (5mg/tablet) was 3mg/m2/day to the maximum dose of 15mg. The dosage ratio was 1:2 and the administration time was 8:00 and 21:00. The initial dose of dexamethasone (0.75mg/tablet) was 0.3mg/m2/day to the maximum dose of 0.75mg and the administration time was 21:00.

The primary objective was to evaluate the effects of different dosage forms of glucocorticoid on the recovery of reproductive function in patients with 21α-hydroxylase deficiency. The primary end point is to evaluate menstrual cycles with ovulation in female patients (including menstrual period, menstrual frequency per year) and sperm count in male patients among the three groups. The secondary endpoint were: 1) The levels of progesterone, 17OHP, testosterone, androstenedione, sex hormone binding protein were measured at follicular phase in female patients and male unlimited in the first month and every three months thereafter; 2) The change of BMI, waist circumference, hip circumference, visceral and subcutaneous fat area, body and liver fat content after one year treatment; 3) The change of blood pressure, fasting blood glucose, fasting insulin, HbA1c, blood lipid profile after one year treatment; 4) The change of bone mineral density after one year; 5) The change of mental health status compared with baseline after one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with 21α-OHD. The reference standard was baseline 17OHP (in the morning of follicular phase in female patients, men unlimited) or after cosyntropin stiimulation > 10ng/ml;
2. Age: >14 years old;
3. Post-puberty;

Exclusion Criteria:

1. Other diseases present with adrenocortical dysfunction, such as primary adrenal hypofunction, Cushing's syndrome, pituitary tumor, etc;
2. Other diseases with hyperandrogenemia were not treated, such as ovarian tumor;
3. Other diseases with HPG axis dysfunction were not treated, such as severe obesity (BMI > 35kg / m2), anorexia nervosa, thyroid dysfunction, etc;
4. Other diseases causing ovarian dysfunction, such as ovarian tumor, endometriosis, primary ovarian failure, etc;
5. History of adrenal and / or pituitary surgery;
6. Elevated AST/ALT (AST > 35 U/L, ALT > 55 U/L)
7. Other diseases need glucocorticoid treatment, such as autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis, autoimmune diseases such as wind dampness heat, rheumatic myocarditis, idiopathic pulmonary fibrosis, autoimmune liver disease, inflammatory bowel disease and amyloidosis, and allergic diseases such as bronchial asthma, exogenous allergic alveolitis and serum diseases, acute urticaria, vascular edema, hematological diseases such as idiopathic thrombocytopenic purpura, immune hemolysis and aplastic anemia, granulocytopenia, other iritis, keratitis, severe drug-induced dermatitis, eczema, etc.
8. Other diseases may lead to the failure of research intervention;
9. Are currently participating in another intervention study or participating in other drug clinical trials within 30 days;
10. No informed consent was signed;
11. According to the researcher's judgment, there is any situation affecting the study compliance;
12. Any other circumstances that are considered by the doctor to be prohibited from participating in the trial.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of ovulatory menstruation in female patients | up to 1 year
The average sperm count in male patients | up to 1 year

SECONDARY OUTCOMES:
The average levels of progesterone | up to 1 year
  Progesterone will be detected at follicular phase (day 2~8) in female patients.
Mean serum concentrations of 17OHP | up to 1 year
Mean serum concentrations of testosterone | up to 1 year
Mean serum concentrations of androstenedione | up to 1 year
Change in BMI | up to 1 year
Change in waist circumference | up to 1 year
Change in blood pressure | up to 1 year
Change in fasting glucose levels | up to 1 year
Change in fasting insulin levels | up to 1 year
Change in 2-hour postprandial glucose levels | up to 1 year
Change in 2-hour postprandial insulin levels | up to 1 year
Change in bone mineral density | up to 1 year
Change in blood metabolomics profile measurement | up to 1 year
  In aid of LC/MS and GC-MS technique, we will measure the metabolomics molecular profile in blood samples before and after treatment. The metabolomics measurement will help to detect the profile of all kinds of hormones, bile acid species, lipids species and amino acid species.
mental health status | up to 1 year
  The Self-reporting inventory ( SCL-90) will be used to evaluate the changes of patients' psychological state at baseline and after one-year treatment from 10 aspects, including somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, terror, paranoia, psychotic and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China